CLINICAL TRIAL: NCT06318468
Title: Exploring the Effectiveness of Utilizing Various Teaching Methods to Enhance the Comprehensive Nursing Assessment Skills of Newly Recruited Nursing Personnel
Brief Title: The Effectiveness of Various Teaching Methods to Enhance the Comprehensive Nursing Assessment Skills of New Nurses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N202306106
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: Competence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Humanoid diagrams training program (Experimental): The experimental group will receive the nursing health assessment teaching for 50 minutes and discussion using humanoid diagrams for 40 minutes to learn comprehensive nursing assessment.
  Interventions: Other: Nursing health assessment teaching and discussion using humanoid diagrams
- comparison group (Active Comparator): The comparison group will receive health assessment teaching for 50 minutes and discussion using case discussion for 40 minutes to learn comprehensive nursing assessment.
  Interventions: Other: Nursing health assessment teaching and discussion using case study

INTERVENTIONS:
Other: Nursing health assessment teaching and discussion using humanoid diagrams — The experimental group will receive the nursing health assessment teaching for 50 minutes and discussion using humanoid diagrams for 40 minutes to learn comprehensive nursing assessment.
  Arms: Humanoid diagrams training program
Other: Nursing health assessment teaching and discussion using case study — The comparison group will receive the nursing health assessment teaching for 50 minutes and discussion using case study for 40 minutes to learn comprehensive nursing assessment.
  Arms: comparison group

SUMMARY:
This study is going to compare different teaching strategies for improving newly recruited nurses' comprehensive nursing assessment skills.

DETAILED DESCRIPTION:
Comprehensive nursing assessment is imperative for newly recruited nursing personnel to holistically identify patients' issues, thereby ensuring the provision of high-quality care. This study employs a randomized controlled trial design and will be conducted at a medical center in northern Taiwan. Eligibility criteria for participation require individuals to be new nurses entering the hospital for the first time and lacking prior clinical work experience. Those working part-time will be excluded from the study. A projected enrollment of 60-80 participants includes 30-40 nurses in both the intervention and comparison groups. Nurses assigned to the intervention group will receive nursing health assessment instruction and engage in discussions utilizing humanoid diagrams. In contrast, nurses in the comparison group will undergo health assessment instruction and discussions using case studies. Questionnaires were administered at baseline, immediately post-intervention, and five weeks thereafter to assess the effects of the two training programs.

ELIGIBILITY:
Inclusion Criteria:

* nurses who enter the hospital for the first time
* nurses have not yet gained clinical work experience

Exclusion Criteria:

* nurses who work in part-time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive health assessment questionnaire | Baseline, before the intervention(T0)
  It is a questionnaire that measures nurses' comprehensive health assessment competency.
Comprehensive health assessment questionnaire | Immediately following after the intervention(T1)
  It is a questionnaire that measures nurses' comprehensive health assessment competency.
Comprehensive health assessment questionnaire | Five weeks after the intervention(T2)
  It is a questionnaire that measures nurses' comprehensive health assessment competency.
Confidence scale (C-scale) | Baseline, before the intervention(T0)
  It is a scale designed to measure participants' confidence in performing the comprehensive nursing assessment.
Confidence scale (C-scale) | Immediately following after the intervention(T1)
  It is a scale designed to measure participants' confidence in performing the comprehensive nursing assessment.
Confidence scale (C-scale) | Five weeks after the intervention(T2)
  It is a scale designed to measure participants' confidence in performing the comprehensive nursing assessment.

SECONDARY OUTCOMES:
Course satisfaction questionnaire | Immediately following after the intervention(T1)
  The scale is designed to measure participants' level of satisfaction with the teaching methods.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Fen Tang, MSN, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (2):
- Taiwan (2):
  - Taipei Municipal Wan Fang Hospital-commissioned by Taipei Medical University / Taipei Taiwan, Taipei
  - Taipei Medical University WanFang Hospital, Taipei